CLINICAL TRIAL: NCT02872766
Title: A Pilot Evaluation of the Safety and Efficacy of Topographically Customized Corneal Cross Linking for the Treatment of Myopia.
Brief Title: Evaluation of the Safety and Efficacy of Corneal Cross Linking for the Treatment of Myopia.
Acronym: CXLMyopie
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15 7714 03
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Corneal cross linking (CXL) (Experimental): Applying riboflavin 0,22% to 0,25 % up to 20 minutes . Then, the eyes are exposed to Ultraviolet A light with the KXL II system according to the programmed treatment pattern.
  Interventions: Device: CXL Myopia

INTERVENTIONS:
Device: CXL Myopia — Applying riboflavin 0,22% to 0,25 % up to 20 minutes . Then, the eyes are exposed to UVA light with the KXL II system according to the programmed treatment pattern.

SUMMARY:
43 Subjects (43 eyes) qualified for participation will undergo the required screening procedures to determine study eligibility. The surgical protocol involves applying riboflavin 0,22% to 0,25 % up to 20 minutes . Then, the eyes will be exposed to UVA (ultraviolet A) light with the KXL II system according to the programmed treatment pattern.

All use of the KXL II system will be in accordance with the general instructions in the operator's manual. All subjects will be evaluated at screening, Day 3, and 1, 3, 6 ,12 and 24 months after treatment.

Manual keratometry, manifest refraction, uncorrected visual acuity, best corrected visual acuity, slit lamp biomicroscopy, pentacam measurements and placido disc topography (TMS), will be obtained at baseline and at appropriate times after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Willingness to follow all instructions and comply with schedule for follow up visits
* Having myopia with manifest refraction spherical equivalent of -1.00 to -2.50 D, with cylindrical component pl to -0.75 D
* Social security insurance or equivalent

Exclusion Criteria:

* sensitivity to the use of the test article(s)
* hypersensitivity to local anesthesics
* Corneal pachymetry that is < 480 microns
* Eyes with keratoconus
* Eyes which are aphakic or with corneal intacs
* Previous ocular condition (other than refractive error) in the eye to be treated that may predispose the eye for future complications. For example: History of corneal disease (e.g., herpes simplex, recurrent erosion syndrome, corneal dystrophy, refractive keratotomy etc.), clinically significant corneal scarring in the crosslinking treatment zone
* Pregnancy or lactation
* Patients with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing
* Taking Vitamin C (ascorbic acid) supplements within 1 week of the cross-linking treatment.
* Juridical protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 1 month
Best corrected visual acuity | 3 months
Best corrected visual acuity | 6 months
Best corrected visual acuity | 12 months
Best corrected visual acuity | 24 months

SECONDARY OUTCOMES:
Adverse events | 1 month
  Clinical examination and slit lamp biomicroscopy
Adverse events | 3 months
  Clinical examination and slit lamp biomicroscopy
Adverse events | 6 months
  Clinical examination and slit lamp biomicroscopy
Adverse events | 12 months
  Clinical examination and slit lamp biomicroscopy
Adverse events | 24 months
  Clinical examination and slit lamp biomicroscopy
Uncorrected visual acuity | 3 months
Mean change in manifest refraction spherical equivalent from baseline | 3 months
Mean change in corneal curvature from baseline | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: François MALECAZE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No